CLINICAL TRIAL: NCT01987687
Title: Effect of Timing of a Post-exercise Oral Glucose Tolerance Test on Glycaemic Control.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, PhD, Research Fellow, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 32W7; 32W7
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Area Under Curve [N06.850.520.830.200]
MeSH Terms: interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rest (Active Comparator): Breakfast followed by a rest period prior to OGTT.
  Interventions: Behavioral: Rest
- Exercise-immediate (Experimental): Breakfast followed by exercise and an immediate OGTT
  Interventions: Behavioral: Exercise
- Exercise-delay (Experimental): Breakfast followed by exercise and a delayed (1 h) OGTT.
  Interventions: Behavioral: Exercise; Behavioral: Delay

INTERVENTIONS:
Behavioral: Exercise — Exercise at 55% of maximum power output for 30 min.
  Arms: Exercise-delay; Exercise-immediate
Behavioral: Rest — Rest for 30 min
  Arms: Rest
Behavioral: Delay — Delay between exercise and OGTT
  Arms: Exercise-delay

SUMMARY:
Postprandial glycaemic control is an important risk factor for the development of type 2 diabetes, cardiovascular disease and all-cause mortality.

Previous research has demonstrated that exercise performed in the postprandial state paradoxically results in a deterioration in glucose tolerance in the immediate post-exercise period (Gonzalez et a. 2013; Gonzalez and Stevenson 2013). This study aims to assess the timecourse of this post-exercise effect.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (18-25 kg/m2)
* Physically active (>or= 3 times per week)
* Male

Exclusion Criteria:

* Contraindications to exercise
* Food intolerances
* Food allergies

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-02 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Postprandial glucose concentration area under the curve | 90 min
  Blood glucose concentrations will be sampled every 15 min following an oral glucose tolerance test.

SECONDARY OUTCOMES:
Postprandial insulin concentration area under the curve | 90 min
  Insulin concentrations will be determine every 15 min following an oral glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Javier T Gonzalez, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Background] Gonzalez JT, Stevenson EJ. Assessment of the post-exercise glycemic response to food: considering prior nutritional status. Nutrition. 2014 Jan;30(1):122-3. doi: 10.1016/j.nut.2013.05.015. Epub 2013 Sep 18. No abstract available. PMID 24054351
- [Background] Gonzalez JT, Veasey RC, Rumbold PL, Stevenson EJ. Breakfast and exercise contingently affect postprandial metabolism and energy balance in physically active males. Br J Nutr. 2013 Aug;110(4):721-32. doi: 10.1017/S0007114512005582. Epub 2013 Jan 29. PMID 23340006